CLINICAL TRIAL: NCT01974518
Title: A PILOT STUDY TO ASSESS THE EFFICACY OF RITUXIMAB VERSUS COMBINATION OF RITUXIMAB AND INTRAVENOUS CYCLOPHOSPHAMIDE IN THE TREATMENT OF REFRACTORY PEMPHIGUS
Brief Title: Comparative Study of Rituximab Versus Combination of Rituximab and Intravenous Cyclophosphamide in Severe Pemphigus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uprety Shraddha (Unknown)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Sponsor-Investigator, Uprety Shraddha, Junior Resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9187-PG-2012
Record Dates: First submitted 2013-10-04; First posted 2013-11-01 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Pemphigus
Keywords: Pemphigus; Rituximab; Rituximab and IV cyclophosphamide combination; B cell re-population characteristics following Rituximab
MeSH Terms: conditions — Pemphigus | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab (Active Comparator): Inj Rituximab 1 gram IV given on day 0 and day 15
  Interventions: Drug: Rituximab and Cyclophosphamide IV
- Combination of Rituximab and Cyclophosphamide IV (Active Comparator): IV Rituximab 1gram on day 0 and 15 750 mg IV cyclophosphamide in 250 ml of NS over 2-3 hr on day 1 and day 16
  Interventions: Drug: Rituximab and Cyclophosphamide IV

INTERVENTIONS:
Drug: Rituximab and Cyclophosphamide IV

SUMMARY:
The purpose of this study is to compare the effectiveness of rituximab alone vs combination of rituximab and cyclophosphamide in the treatment of pemphigus not responding adequately to routine medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of pemphigus based on clinical, histopathological and immunological features the following:
* Refractory disease defined as continuing extension of old lesions, development of new lesion, or failure of established lesions to begin to heal despite 3 weeks of therapy on 1.5 mg/kg/day of prednisolone or its equivalent with or without the concurrent use of cyclophosphamide 2mg/kg/day for 12 weeks or azathioprine 2.5 mg/kg/day for 12 weeks. Patients who fail to respond to 6 DCP/DP are also considered as refractory disease.

Exclusion Criteria:

* Infections- Hepatitis B, Hepatitis C, HIV, active tuberculosis or sepsis.
* Abnormal liver function tests and renal function tests
* Known cardiac arrhythmia or conduction abnormality
* Systolic ejection fraction <40%
* Pregnancy and breast feeding
* Severely decreased bone marrow functions.
* Known history of bladder cancer or hemorrhagic cystitis
* Known allergy to cyclophosphamide
* Patients of reproductive age group who haven't completed their family
* Known hypersensitivity to murine proteins.
* Patients who do not consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Study the clinical efficacy of IV rituximab vs IV rituximab and IV cyclophosphamide combination for treatment of refractory pemphigus in terms of early and late end points as defined by the international pemphigus committee | upto 9 months
  Primary outcome measures being
  1. Time taken for control of disease activity
  2. Time taken for achievement of partial remission
  3. Time taken for achievement of complete remission

SECONDARY OUTCOMES:
Study the characteristics of B cell depletion and repopulation following IV rituximab and combination of IV cyclophosphamide with IV rituximab. | upto 9 months
  Flowcytometric analysis of CD19+ve27-ve naïve B cells count, CD19+ve27+ve memory B cells count and CD24highCD38high transitional cell count will be performed at baseline, 3rd month, 6th month and 9th month.

OTHER OUTCOMES:
To study the difference in relapse rate | upto 9 months
to study the total cumulative dose of corticosteroids adminstered and adjuvants required among patients of the 2 treatment groups | upto 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Shraddha Uprety, MBBS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (2):
- India (2):
  - PGIMER, Chandigarh, Chandigarh
  - Post-graduate Institute of Medical Education and Research, Chandigarh, Chandigarh